CLINICAL TRIAL: NCT00599274
Title: A Multicenter, Prospective and Retrospective, Long-Term Observational Study of AVONEX® and Rebif® to Determine the Efficacy, Tolerability, and Safety in Subjects With Relapsing Multiple Sclerosis (MS)
Brief Title: Study to Determine if Avonex and Rebif Work Comparably Well in Subjects With Relapsing Multiple Sclerosis
Acronym: PROOF
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Other Study IDs: C-862
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Interferon beta 1a; Avonex
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: This group was treated with Avonex once a week
  Interventions: Drug: Interferon beta-1a
- B: This group was treated with Rebif three times a week
  Interventions: Drug: Interferon beta-1a

INTERVENTIONS:
Drug: Interferon beta-1a — injection once a week
  Other Names: Avonex
  Groups: A
Drug: Interferon beta-1a — injection three times a week
  Other Names: Rebif
  Groups: B

SUMMARY:
The purpose of this study is to find out if weekly Avonex works as well as three times a week Rebif in subjects with relapsing multiple sclerosis.

DETAILED DESCRIPTION:
This is a Phase 4, multicenter, prospective and retrospective, long-term observational study of Avonex® and Rebif® to determine the efficacy, tolerability, and safety in subjects with relapsing MS.

ELIGIBILITY:
Inclusion Criteria:

* Must have been receiving AVONEX® or Rebif®.
* Must have a confirmed diagnosis of relapsing-remitting MS using the Poser criteria.
* Must have experienced at least 2 relapses within the 3 year period prior to the initiation of treatment.
* Must have an EDSS score of 0.0 to 5.5, inclusive.

Exclusion Criteria:

* History of severe allergic or anaphylactic reaction or hypersensitivity to human albumin, to any interferon, or to other components of the drug formulation.
* History of poorly controlled hypertension and/or other clinically significant major disease.
* History of uncontrolled seizures within the 3 months prior to enrollment.
* History of suicidal ideation or an episode of severe depression within the 3 months prior to enrollment.
* Serious local infection or systemic infection within 8 weeks prior to enrollment.
* Treatment with certain other agents to treat MS symptoms or underlying disease.
* Treatment with any investigational product
* Previous participation in this study.
* Other Protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: subjects with relapsing remitting Multiple Sclerosis taking AVONEX® or Rebif®.
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2002-08; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Investigator, Principal Investigator — Biogen
Locations (11):
- United States (8):
  - Research Site, Los Angeles, California
  - Research Site, Walnut Creek, California
  - Research Site, Shreveport, Louisiana
  - Research Site, Worcester, Massachusetts
  - Research Site, Charlotte, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Edmonds, Washington
  - Research Site, Milwaukee, Wisconsin
- Coordinating Research Site, Woodville, Australia
- Coordinating Research Site, Linz, Austria
- Coordinating Research Site, Halifax, Nova Scotia, Canada